CLINICAL TRIAL: NCT01622530
Title: Development of a Simulation Tool for Upper Extremity Prostheses
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Stephanie L. Carey, Assistant Research Professor, University of South Florida
Other Study IDs: Pro00000991; 09128006 (Other Grant/Funding Number: U.S. Department of Defense (TATRC))
Record Dates: First submitted 2012-06-07; First posted 2012-06-19 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Traumatic Amputation of Upper Limb, Level Unspecified

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Amputees: upper limb amputees
- Non-amputees: No longer recruiting non-amputees

SUMMARY:
Amputees often choose not to wear prostheses due to marginal performance or may settle for a prosthesis that offers only cosmetic improvement, but lacks function. A simulation tool consisting of a robotics-based human body model (RHBM) to predict functional motions, and integrated modules for aid in prescription, training, comparative study, and determination of design parameters of upper extremity prostheses will be developed.

The main objective of collecting and analyzing human movement during several common tasks is to optimize and validate the robotics based human model. The range of motion data of subjects performing activities of daily living such as opening a door, turning a wheel, grooming, eating, bilateral lifting, as well as recreational and sport activities such as swinging a baseball bat, and golf club will be analyzed. This motion analysis data will also be used to compare data between four groups: a control group (n=10), a braced group simulating prosthesis use (n=10), a group wearing a transradial prosthesis (n=10) and a group wearing a transhumeral prosthesis (n =10).

DETAILED DESCRIPTION:
Data will be collected by an 8 camera Vicon© motion analysis system during one 3-4 hour testing period. Forty-five reflective markers will be attached to subjects skin and clothing via a double sided adhesive electrode collar. The cameras work on an infrared spectrum and the markers are passive reflective spheres. Relations between marker positions and anatomical / known positions on the body are used to calculate the positions of body segments.This analysis will provide information on movement strategies, compensatory motion, and socket movement associated with the selected tasks for transradial and transhumeral prostheses. Differences in the range of motion of the prostheses users and control subjects will be calculated to determine compensatory motion. The movement of the prosthesis's socket as a function of task and other factors will also be measured. Measured data will be used to minimize error in the simulation of the upper body movement. Knowledge of human motor function given in the recorded data can be extended to give insight to movement parameters when designing new prosthetics. Simulations will be optimized to the collected data using a regressive best fit method.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be capable of providing an informed consent.
* Normal healthy adult subjects and upper limb amputees that currently use a prosthesis to complete activities of daily living will be included.

Exclusion Criteria:

* Subjects younger than 18 or older than 65 will be excluded.
* Adults that are unable to consent will be excluded from the study.
* Subjects that have health issues or injuries that would prevent them from lifting five pounds or completing simple tasks of daily living will be excluded from the study.
* Subjects will be asked if they are able to lift five pounds, open a door and drink from a cup without pain or injury. Before study set up and recording begins, subjects will be asked to practice these tasks to insure that they are capable of completing them.
* Pregnant women will be excluded from this study due to the changes in some physical abilities during pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups will be studied: non-amputees and upper limb amputees. The subjects will be recruited from around the community.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Shoulder angle | During task completion
  The shoulder angle (rotation, flexion/extension and abduction/adduction) will be measured during several tasks during one 3-4 hour testing period.
Elbow angle | During task completion
  The elbow angle ( flexion/extension and forearm pronation/supination) will be measured during several tasks during one 3-4 hour testing period.
Wrist angle | During task completion
  The wrist angle (flexion/extension and abduction/adduction) will be measured during several tasks during one 3-4 hour testing period.
Torso angle | During task completion
  The torso angle (rotation, forward/backward bending and right/left sideways bending) will be measured during several tasks during one 3-4 hour testing period.

SECONDARY OUTCOMES:
Validation of robotics based human body model | After motion data analysis
  The robotics based human body model will be validated by comparing the joints (shoulder, elbow, wrist, torso) angles collected from the motion analysis system while participants are completing activities of daily living with the joint angles predicted by the model. The two data sets will be compared using a root mean error calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Dubey, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Floria RRT building, Tampa, Florida, United States

REFERENCES:
- See also: Center for Rehabilitation, Robotics and Assistive Technologies — http://carrt.eng.usf.edu